CLINICAL TRIAL: NCT07040397
Title: Comparing an Electronic Approach to the Human Massage Therapist.
Brief Title: Electronic Approach to the Human Massage Therapist
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael R. Mueller, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-002863
Record Dates: First submitted 2025-06-05; First posted 2025-06-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lower Back Pain
Keywords: massage; Low Back Pain; automated massage; EMMA (expert manipulative massage automation); electric massager
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: 20 will be randomized to EMMA and 20 to a certified massage therapist. Everyone will receive a massage treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Indirect person massage therapy (Experimental): A massage therapist will program and direct an Artificial Intelligence Robotic Arm (EMMA) to deliver massage therapy. EMMA executes massages through soft treatment modules that are warmed to a temperature of between 38℃ and 40℃ to mimic human touch. This treatment will last approximately 20 minutes.
  Interventions: Device: EMMA massage therapy
- Direct person massage therapy (Active Comparator): Clinical massage treatment procedures are delivered by a clinically licensed massage therapist. This treatment will last approximately 20 minutes.
  Interventions: Other: Clinical massage treatment

INTERVENTIONS:
Device: EMMA massage therapy — Expert Manipulative Massage Automation (EMMA) is equipped with sensors to measure muscle stiffness and uses 3D vision technology to measure muscle stiffness and identify pressure points while delivering a massage to patients. Following that, the electronic massager will determine the best course of action for our patients based on the information stored by our Artificial Intelligence and EMMA's robotic arm will perform the massage. EMMA executes massages through soft treatment modules that are warmed to a temperature of between 38℃ and 40℃ to mimic human touch.
  Arms: Indirect person massage therapy
Other: Clinical massage treatment — The direct person clinical massage treatment will be delivered by a clinical licensed massage therapist. The type of massage will follow the EMMA massage in that it will be a deep tissue massage (to mimic the Tuina massage) and generally will be for about 30 minutes to once again mimic the duration of massage therapy of the EMMA.
  Arms: Direct person massage therapy

SUMMARY:
The purpose of this study is to gather information about patient experience receiving a massage through a robotic EMMA (Expert Manipulative Massage Automation) compared to receiving a massage from a massage therapist.

DETAILED DESCRIPTION:
Patients being evaluated in an outpatient service will be invited to participate in this study if they report a primary pain point in Low Back. Once they are enrolled in the study, they will be randomized to the type of massage therapy they will receive. Direct massage therapy through a certified massage therapist or indirect massage therapy through EMMA operated by a certified massage therapist.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age or older.
* report a primary pain point in the lower back.
* Pain intensity reported at baseline
* Women of childbearing potential who self-report not being pregnant and agree to employ an effective method of birth control (surgical sterilization or oral contraceptives, barrier method with spermicides, intrauterine device, etc.) during the study period
* be able to participate fully in all aspects of the study.
* have understood and signed study informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients with the inability to stay in a prone position
* Patients with bleeding disorders
* Patients with allergies and/or local skin affectations
* have used pain medications or participated in a pain treatment within three days of study enrollment.
* have an implanted device (including a lap band) in the targeted area of massage therapy.
* have used an investigational drug within 30 days of study enrollment.
* have a history of any major cardiovascular events including heart valve disease, ongoing angina, cardiac arrhythmias, congestive heart failure, acute coronary syndrome, stroke, transient ischemic attack, or peripheral vascular disease.
* have clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, lymphatic, respiratory, metabolic disease (such as uncontrolled diabetes type 2) active cancer, actively receiving treatment for cancer or within 1 year of cancer remission.
* surgical intervention for pain within 1 month prior to enrollment.
* active infection, wound or other external trauma to the areas to be treated with massage therapy.
* have a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled | baseline to end of study (year 2)
  Feasibility will be determined by the total number of patients screened in order to accrue the 40 needed to complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mueller, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20582560